CLINICAL TRIAL: NCT07299383
Title: Comparison of Local Anesthesia With the Fully Awake Tourniquet-Free Local Anesthesia Technique (WALANT) in Central Venous Catheter Insertion Procedure
Brief Title: WALANT Versus Local Anesthesia in Central Venous Catheter Insertion
Acronym: WALANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ümit arslan, PROFESSOR, Ataturk University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/830; Ayça ÇALBAY (Other: Atatürk University)
Record Dates: First submitted 2025-11-26; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Trauma (Including Fractures); Dialysis Catheter; Malnutrition Severe
Keywords: walant; cenral venous catheter; local anesthesia; lidocain; epinephrine
MeSH Terms: conditions — Wounds and Injuries | interventions — Anesthesia, Local; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Active Comparator): After selecting the area where the CVC would be inserted (femoral vein, subclavian vein, jugular vein), anatomical localization was determined without using any guide such as USG, and the vein where the procedure would be performed was determined by using a 10cc syringe with negative pressure and passing through the skin and subcutaneous tissues. An average of 2-10ml of WALANT solution was injected into the designated 3x3cm area while the needle tip was slowly withdrawn. After waiting 20 minutes, CVC placement was performed. Patient assessments were recorded using a visual analog scale before and at the end of the procedure.
  Interventions: Procedure: local anesthesia with walant solution; Procedure: Local anesthesia with lidocaine
- Control (Lidocaine group) (Active Comparator): For the control group, patients requiring a CVC were selected as single-blind and underwent the procedure in the emergency resuscitation room. After selecting the catheter insertion site after marking the anatomical location, the vein to be treated was identified by using a 10cc syringe and applying negative pressure to the skin and subcutaneous tissues. While the needle was slowly withdrawn, local anesthesia was induced by applying an average of 2-10ml lidocaine (1.5-2 mg/kg) to the designated 3x3cm area. CVC insertion was then performed according to routine procedures. Patient assessments were recorded before and after the procedure using a VAS.
  Interventions: Procedure: Local anesthesia with lidocaine

INTERVENTIONS:
Procedure: local anesthesia with walant solution — Walant solution was prepared using 5 ml lidocaine, 4 ml 0.9% isotonic, 1 ml 8.5% sodium bicarbonate, 1 ml 1/1000 epinephrine and an average of 2-10 ml of WALANT solution was injected into a 3x3 cm area
  Arms: Case group
Procedure: Local anesthesia with lidocaine — ocal anesthesia was induced by applying an average of 2-10ml lidocaine (1.5-2 mg/kg) to the designated 3x3cm area. CVC insertion was then performed according to routine procedures.

SUMMARY:
The goal of this clinical trial is to find out whether WALANT is an alternative local anesthesia method that can increase patient comfort and reduce pain during CVC procedure, which is one of the invasive procedures to be performed especially in areas where bleeding control is difficult.

The main questions it aims to answer are:

* Can we offer an alternative local anesthesia method that can be used to treat patients who require CVC insertion with minimum pain and maximum comfort?
* Can the WALANT technique reduce the risk of complications during CVC insertion?

Participants were:

randomized using a single-blind allocation method based on hospital file numbers: odd numbers received WALANT and even numbers received lidocaine. The WALANT solution was prepared according to the standard protocol and injected into a 3×3 cm target area 20 minutes before catheter insertion. CVCs were placed without ultrasound guidance in jugular, subclavian, or femoral veins by anatomical localization. Pain intensity was assessed using the Visual Analog Scale (VAS) before and after the procedure. In the control group, after marking the anatomical location, the vein where the procedure would be performed was identified by using a 10cc syringe, which was then passed through the skin and subcutaneous tissues using negative pressure. As the needle tip was slowly withdrawn, local anesthesia was induced with an average of 2-10ml lidocaine (1.5-2 mg/kg) applied to the designated 3x3cm area. The CVC was then placed according to routine procedures. Patient assessments were recorded using a visual analog scale before and after the procedure.

DETAILED DESCRIPTION:
Patients were included in the study if they were older than 18 years, non-pregnant, had a Glasgow Coma Scale score of 15, were oriented and cooperative, and had a hemorrhagic shock stage of at most 1 or were not in hemorrhagic shock. Patients were excluded if they were younger than 18 years, pregnant, had a Glasgow Coma Scale score of <15, were unoriented and cooperative, were in hemorrhagic shock stage >1, had coagulopathy, increased intracranial pressure, target vessel hemorrhage, obstruction, or thrombus, skin infection in the relevant area, or had burns. Sixty-four patients were included in the study between the targeted dates. Patient epidemiological characteristics, the vessel from which CVC was administered, pre- and post-treatment VAS scores, chronic diseases, medications, and any complications were recorded in the prepared case forms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are over 18 years of age, not pregnant, have a Glasgow Coma Scale score of 15, are oriented and cooperative, and have a hemorrhagic shock stage of at most 1 or are not in hemorrhagic shock.

Exclusion Criteria:

* Patients who are younger than 18 years of age, pregnant, have <15 points on the Glasgow Coma Scale, are not oriented or cooperative, are in hemorrhagic shock stage >1, have coagulopathy, increased intracranial pressure, bleeding-obstruction-thrombus in the target vessel, skin infection in the relevant area, or have burns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the pain felt by patients after central venous catheter placement when local anesthesia is performed with Lidocaine and when it is performed with the Wide Awake Tourniquet-Free Local Anesthesia Technique (WALANT). | 45 minutes for each patient.
  To measure pain, participants were asked to describe the pain felt before and after central venous catheter insertion using a VISUAL ANALOG SCALE (VAS). They were asked to give a score of 10 for the highest pain felt and 0 for the situation where they felt no pain.
Comparison of Pain Experienced by Patients After Central Venous Catheter Insertion Procedure with Local Anesthesia with Lidocaine and the Wide-Awake Tourniquet-Free Local Anesthesia Technique (WALANT) | The time from the beginning of the CVC insertion process until the patient can describe the pain he/she feels is a maximum of 30 minutes. The study duration was 45 minutes per patient.
  To measure pain, patients were asked to describe the pain felt before and after central venous catheter insertion using a VISUAL ANALOG SCALE (VAS). They were asked to give a score of 10 for the highest pain experienced and 0 for no pain at all. A Visual Analogue Scale (VAS) is one of the pain rating scales used for the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. From the patient's perspective, this spectrum appears continuous; their pain does not take discrete jumps, as a categorization of none, mild, moderate and severe would suggest.
Pain felt after local anesthesia | The maximum time elapsed from the moment the patient was able to describe the pain felt after the local anesthesia procedure was 30 minutes.
  To measure pain, patients were asked to describe the pain felt before and after central venous catheter insertion using a VISUAL ANALOGUE SCALE (VAS). They were asked to give a score of 10 for the highest pain experienced and 0 for no pain at all.

CONTACTS AND LOCATIONS:
Overall Officials: SULTAN TUNA AKGÖL GÜR, ASSOCIATE PROFESSOR, Principal Investigator — ATATÜRK UNİVERSİTY; MURAT MAKSUT ÇALBAY, SPECİALİST, Principal Investigator — ERZURUM CİTY HOSPİTAL; MUHAMMED ÇAĞRI AYKUT, MD, Principal Investigator — ATATÜRK UNİVERSİTY; ORHAN ENES TUNÇEZ, MD, Principal Investigator — AMASYA SULUOVA STATE HOSPITAL
Locations (1):
- Atatürk University Research Hospital, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Epidemiological data in the case form prepared for the study, chronic disease/chronic medication use, VAS values of the study, and data on the presence of complications can be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The desired data can be shared within 2 years after the study is completed and published (excluding patients' personal data).
Access Criteria: Individuals with at least a medical doctor's degree who are mentors on topics related to the study, planning a similar study design, or planning a course or academic presentation on this topic are eligible to access the data.
  The Correponder Author can be contacted for data sharing.
  Email is preferred for communication.
URL: https://avesis.atauni.edu.tr/researcher

REFERENCES:
- [Result] Arik HO, Coskun T, Kose O. Management of spaghetti wrist under WALANT technique. Hand Surg Rehabil. 2021 Oct;40(5):655-659. doi: 10.1016/j.hansur.2021.06.006. Epub 2021 Jun 21. PMID 34166849
- [Result] Abell RG, Page IH. THE REACTION OF PERIPHERAL BLOOD VESSELS TO ANGIOTONIN, RENIN, AND OTHER PRESSOR AGENTS. J Exp Med. 1942 Mar 1;75(3):305-14. doi: 10.1084/jem.75.3.305. PMID 19871185
- [Result] Yayla EM, Ozdemir L. Effect of Inhalation Aromatherapy on Procedural Pain and Anxiety After Needle Insertion Into an Implantable Central Venous Port Catheter: A Quasi-Randomized Controlled Pilot Study. Cancer Nurs. 2019 Jan/Feb;42(1):35-41. doi: 10.1097/NCC.0000000000000551. PMID 29199999
- [Result] Samantaray A, Hanumantha Rao M, Sahu CR. Additional Analgesia for Central Venous Catheter Insertion: A Placebo Controlled Randomized Trial of Dexmedetomidine and Fentanyl. Crit Care Res Pract. 2016;2016:9062658. doi: 10.1155/2016/9062658. Epub 2016 Apr 21. PMID 27200187
- [Result] Dar QA, Avoricani A, Rompala A, Levy KH, Shah NV, Choueka D, White CM, Koehler SM. WALANT Hand Surgery Does Not Require Postoperative Opioid Pain Management. Plast Reconstr Surg. 2021 Jul 1;148(1):121-130. doi: 10.1097/PRS.0000000000008053. PMID 34181608
- [Result] Moscato L, Laborde A, Kouyoumdjian P, Coulomb R, Mares O. Trapeziometacarpal (TMC) arthroplasty under Wide Awake Local Anesthesia with No Tourniquet (WALANT) versus Local Anesthesia with peripheral nerve blocks (LAPNV): Perioperative pain and early functional results in 30 patients. Hand Surg Rehabil. 2021 Sep;40(4):453-457. doi: 10.1016/j.hansur.2021.03.006. Epub 2021 Mar 26. PMID 33775887
- [Result] Tahir M, Chaudhry EA, Zaffar Z, Anwar K, Mamoon MAH, Ahmad M, Jamali AR, Mehboob G. Fixation of distal radius fractures using wide-awake local anaesthesia with no tourniquet (WALANT) technique: A randomized control trial of a cost-effective and resource-friendly procedure. Bone Joint Res. 2020 Jul 1;9(7):429-439. doi: 10.1302/2046-3758.97.BJR-2019-0315.R1. eCollection 2020 Jul. PMID 32905335
- [Result] Wellington I, Cusano A, Ferreira JV, Parrino A. WALANT Technique versus Sedation for Endoscopic Carpal Tunnel Release. Hand (N Y). 2023 Mar;18(2):214-221. doi: 10.1177/15589447211003180. Epub 2021 Apr 9. PMID 33834864
- [Result] Lalonde DH. Conceptual origins, current practice, and views of wide awake hand surgery. J Hand Surg Eur Vol. 2017 Nov;42(9):886-895. doi: 10.1177/1753193417728427. Epub 2017 Sep 8. PMID 28886668
- See also: Ethical files and applications for the study were made through the university system. — https://atauni.edu.tr/
- Available data/document: Study Protocol: AYÇA ÇALBAY — https://atauni.edu.tr/ — online access is not available, accessible via e-mail

DOCUMENTS (3):
  • Study Protocol (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT07299383/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT07299383/SAP_001.pdf
  • Informed Consent Form (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT07299383/ICF_002.pdf